CLINICAL TRIAL: NCT03870139
Title: Effects of Peripheral and Cerebral Electrical Stimulation on Maximal Isometric Strength of Knee Extensors
Brief Title: Cerebral and Peripheral Electrical Stimulation on Isometric Quadriceps Strength
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Assistant Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and knee strength
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cerebral stimulation (Active Comparator): Active transcranial direct current stimulation
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the dominant lower limb) and supraorbital cathode (ipsilateral to the dominant lower limb).
  Interventions: Device: Cerebral stimulation
- Combined stimulation 1 (Experimental): Active peripheral electrical stimulation (PES_sensorial) combined with active transcranial direct current stimulation
  tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  PES_sensorial: 20 minutes, 10Hz (frequency), 100µs (pulse duration), intensity at sensorial level.
  Interventions: Device: Cerebral stimulation; Device: Peripheral stimulation
- Peripheral stimulation (Active Comparator): Active peripheral electrical stimulation (PES_motor).
  PES: 15 minutes, 30Hz (frequency), 100µs (pulse duration), intensity at motor level.
  Interventions: Device: Peripheral stimulation
- Combined stimulation 2 (Experimental): Active sensorial peripheral electrical stimulation (PES_sensorial) combined with active motor peripheral electrical stimulation (PES_motor)
  PES_sensorial: 20 minutes, 10Hz (frequency), 100µs (pulse duration), intensity at sensorial level
  PES_motor: 15 minutes, 30Hz (frequency), 100µs (pulse duration), intensity at motor level.
  Interventions: Device: Cerebral stimulation; Device: Peripheral stimulation

INTERVENTIONS:
Device: Cerebral stimulation — Transcranial direct current stimulation (tDCS) is a noninvasive brain stimulation (NIBS) technique that has been investigated for the management of various health conditions. However, its ergogenic effect still has controversial results.
  Other Names: Transcranial direct current stimulation
  Arms: Cerebral stimulation; Combined stimulation 1; Combined stimulation 2
Device: Peripheral stimulation — Peripheral electrical stimulation (PES) activates a complex neural network involving a series of neurotransmitters and receptors capable of promoting segmental and extrasegmental analgesia. Moreover, recent evidence has shown that PES can activate brain motor areas such as primary motor cortex.
  Arms: Combined stimulation 1; Combined stimulation 2; Peripheral stimulation

SUMMARY:
Quadriceps muscle strength is a key goal to be achieved in rehabilitation protocols for a variety of musculoskeletal conditions. Both cerebral and peripheral electrical stimulations can modulate motor brain areas involved in motor functions and has the potential to optimize muscle capacity. However, their effects on quadriceps function are lacking.

This study aims to investigate the effects of transcranial direct current stimulation (tDCS) and peripheral electrical stimulation (PES) on quadriceps strength in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no complaints of pain, discomfort in the musculoskeletal system.

Exclusion Criteria:

* Musculoskeletal or neurological disorder
* Under medication

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Isometric quadriceps strength | Pre and Post-test (immediately after tDCS)
  Maximal isometric voluntary contraction (Kgf)

SECONDARY OUTCOMES:
Isometric quadriceps strength | During stimulation
  Maximal isometric voluntary contraction (Kgf)
Isometric quadriceps strength | 10 minutes post-stimulation
  Maximal isometric voluntary contraction (Kgf)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No